CLINICAL TRIAL: NCT02275156
Title: Phase 1, Open-label, Single-dose Study of Evolocumab (AMG 145) Administered Subcutaneously to Subjects With Normal Renal Function or Severe Renal Impairment or End Stage Renal Disease Receiving Hemodialysis
Brief Title: Estimation Study to Assess the Effect of Severe Renal Impairment and End-stage Renal Disease Hemodialysis on the Pharmacokinetics of Evolocumab
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140213
Record Dates: First submitted 2014-07-15; First posted 2014-10-27 (Estimated); Results first posted 2016-01-29 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Hyperlipidemia; Mixed Dyslipidemia
Keywords: Subjects with normal renal function or severe renal impairment (RI) or end stage renal disease (ESRD) receiving hemodialysis
MeSH Terms: conditions — Hyperlipidemias; Renal Insufficiency; Kidney Failure, Chronic | interventions — evolocumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evolocumab (Experimental): Participants received a single 140 mg dose of evolocumab subcutaneously on Day 1.
  Interventions: Biological: Evolocumab

INTERVENTIONS:
Biological: Evolocumab — Administered by subcutaneous injection
  Other Names: AMG 145; Repatha

SUMMARY:
The primary objective of this study was to evaluate the pharmacokinetics of evolocumab after a single 140 mg subcutaneous (SC) dose in aduts with normal renal function or severe renal impairment or end-stage renal disease (ESRD) receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of ≥ 18 and ≤ 35 kg/m² at screening.
* Subjects will have low-density lipoprotein cholesterol (LDL-C) of 70-190 mg/dL (inclusive) and on statin therapy.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Subject with current or prior history of statin intolerance
* Subject has previously received Evolocumab (AMG 145) or any other investigational therapy directed against PCSK9
* Known substance abuse (eg, alcohol, licit or illicit drugs) within 12 months of day -1
* Testing positive for alcohol and/or drugs-of-abuse at screening, day -1, or day 1 (alcohol only)
* History of hypersensitivity or allergic reaction to mammalian-derived drug preparations
* Known sensitivity to any of the active substances or their excipients to be administered during dosing, eg, carboxymethylcellulose
* Other exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2014-12-19 (Actual); Study Completion 2014-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Research Site, Denver, Colorado, United States

REFERENCES:
- [Background] Kasichayanula S, Grover A, Emery MG, Gibbs MA, Somaratne R, Wasserman SM, Gibbs JP. Clinical Pharmacokinetics and Pharmacodynamics of Evolocumab, a PCSK9 Inhibitor. Clin Pharmacokinet. 2018 Jul;57(7):769-779. doi: 10.1007/s40262-017-0620-7. PMID 29353350
- [Background] Lee E, Gibbs JP, Emery MG, Block G, Wasserman SM, Hamilton L, Kasichayanula S, Hanafin P, Somaratne R, Egbuna O. Influence of Renal Function on Evolocumab Exposure, Pharmacodynamics, and Safety. Clin Pharmacol Drug Dev. 2019 Apr;8(3):281-289. doi: 10.1002/cpdd.650. Epub 2019 Jan 24. PMID 30676701
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighteen participants were enrolled at 1 center in the United States. The first participant enrolled on 19 August 2014 and the last participant enrolled on 28 October 2014.
Groups:
- Normal Renal Function: Participants with normal renal function (defined as an estimated glomerular filtration rate [eGFR] ≥ 90 mL/min/1.73 m²) received a single 140 mg dose of evolocumab subcutaneously on Day 1.
- Severe Renal Impairment: Participants with severe renal impairment (defined as eGFR 15 to 29 mL/min/1.73 m²) received a single 140 mg dose of evolocumab subcutaneously on Day 1.
- End Stage Renal Disease: Participants with end-stage renal disease (ESRD) requiring hemodialysis received a single 140 mg dose of evolocumab subcutaneously on Day 1.
Period: Overall Study
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (9.9) | 63.3 (7.8) | 57.0 (8.1) | 57.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 4 | 4 | 3 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Black (or African American) | 1 | 1 | 4 | 6
  White | 5 | 5 | 2 | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Serum Concentration (Cmax) of Evolocumab
Description: Serum concentrations of evolocumab were measured by a validated enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) of the assay was 800 ng/mL.
Time Frame: Predose and 4 hours, 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 50 and 57 days postdose
Population: Pharmacokinetic (PK) analysis set (all participants for whom at least 1 PK parameter could be adequately estimated)
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 21.3 (9.00) | 15.1 (8.86) | 11.7 (7.20)

2. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC0-last) for Evolocumab
Time Frame: Predose and 4 hours, 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 50 and 57 days postdose
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
day*μg/mL | 185 (92.5) | 141 (109) | 102 (80.1)

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event was graded using the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4. A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal;
  * life threatening (places the participant at immediate risk of death);
  * requires in patient hospitalization or prolongation of existing hospitalization;
  * results in persistent or significant disability/incapacity;
  * congenital anomaly/birth defect;
  * other medically important serious event.
  The investigator assessed whether each adverse event was possibly related to the study drug.
Time Frame: From the first dose of study drug up until Day 57
Population: Safety analysis set (all participants who received at least 1 dose of study drug)
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
participants
  Any adverse event | 1 | 1 | 2
  Grade ≥ 2 | 1 | 1 | 0
  Grade ≥ 3 | 0 | 1 | 0
  Grade ≥ 4 | 0 | 0 | 0
  Serious adverse events | 0 | 1 | 0
  Leading to discontinuation of study drug | 0 | 0 | 0
  Leading to discontinuation from study | 0 | 0 | 0
  Fatal adverse events | 0 | 0 | 0
  Treatment-related adverse events | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Clinically Relevant Vital Sign or Clinical Laboratory Changes
Description: The investigator reviewed vital signs and laboratory test results and determined whether an abnormal value in an individual participant represented a clinically significant change from the participant's baseline values.
Time Frame: 57 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Anti-evolocumab Antibodies
Description: Blood samples were tested using an electrochemiluminescence-based bridging immunoassay to detect antibodies capable of binding to evolocumab.
Time Frame: 57 days
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
participants | 0 | 0 | 0

6. Secondary Outcome: Area Under the Effect Curve From Baseline to Day 57 (AUECday1-57) for Low-density Lipoprotein Cholesterol (LDL-C)
Description: The derived log-transformed AUECday1-57 for direct LDL-C was analyzed using a mixed-effect analysis of variance model. Log-transformed baseline LDL-C was the covariate.
Time Frame: 4 hours, 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 50 and 57 days postdose
Population: Safety analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL*day
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
mg/dL*day | 4438.6 [3873.3 to 5086.5] | 4087.5 [3555.5 to 4699.1] | 4620.2 [4050.8 to 5269.6]

7. Secondary Outcome: Mean Percent Change From Baseline in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9)
Description: Serum PCSK9 concentrations were determined using a qualified ELISA. The LLOQ of the assay was 15 ng/mL.
  Log-transformed baseline PCSK9 was included in the model as a covariate and participant as a random effect.
Time Frame: Baseline and 4 hours, 2, 3, 4, 6, 8, 11, 15, 22, 29, 43, 50 and 57 days postdose
Population: Safety analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: percent change
Arm/Group | Normal Renal Function | Severe Renal Impairment | End Stage Renal Disease
Number analyzed (Participants) | 6 | 6 | 6
percent change
  Day 1, Hour 4 | -91.69 [-94.66 to -87.09] | -79.20 [-86.63 to -67.64] | -72.95 [-82.59 to -57.97]
  Day 2 | -96.67 [-97.86 to -94.83] | -95.87 [-97.34 to -93.57] | -94.41 [-96.40 to -91.31]
  Day 3 | -96.67 [-97.86 to -94.83] | -96.33 [-97.64 to -94.29] | -95.58 [-97.16 to -93.14]
  Day 4 | -96.67 [-97.86 to -94.83] | -96.33 [-97.64 to -94.29] | -96.53 [-97.77 to -94.61]
  Day 6 | -96.67 [-97.86 to -94.83] | -96.33 [-97.64 to -94.29] | -95.39 [-97.03 to -92.83]
  Day 8 | -96.67 [-97.86 to -94.83] | -96.33 [-97.64 to -94.29] | -95.01 [-96.79 to -92.25]
  Day 11 | -96.67 [-97.86 to -94.83] | -95.96 [-97.40 to -93.71] | -94.69 [-96.58 to -91.75]
  Day 15 | -90.42 [-93.84 to -85.12] | -86.41 [-91.26 to -78.86] | -82.97 [-89.04 to -73.53]
  Day 22 | -65.84 [-78.02 to -46.40] | -57.92 [-72.95 to -34.54] | -60.33 [-74.47 to -38.36]
  Day 29 | -49.12 [-67.26 to -20.93] | -53.66 [-70.21 to -27.91] | -51.88 [-69.03 to -25.23]
  Day 43 | -24.93 [-51.70 to 16.67] | -36.30 [-59.05 to -0.92] | -42.44 [-62.95 to -10.56]
  Day 50 | -2.88 [-37.51 to 50.95] | -26.57 [-52.79 to 14.22] | -37.04 [-59.48 to -2.17]
  Day 57 | -1.46 [-36.60 to 53.14] | -14.49 [-45.03 to 33.02] | -37.74 [-59.93 to -3.25]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up until Day 57
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  Summary of Adverse Events includes only those subjects who received at least one dose of investigational product.
  ESRD = End stage renal disease requiring dialysis.
Groups:
- Evolocumab 140 mg - Normal Renal Function: Participants with normal renal function (defined as an estimated glomerular filtration rate [eGFR] ≥ 90 mL/min/1.73 m²) received a single 140 mg dose of evolocumab subcutaneously on Day 1.
- Evolocumab 140 mg - Severe RI: Participants with severe renal impairment (defined as eGFR 15 to 29 mL/min/1.73 m²) received a single 140 mg dose of evolocumab subcutaneously on Day 1.
- Evolocumab 140 mg - ESRD Requiring Hemodialysis: Participants with end-stage renal disease (ESRD) requiring hemodialysis received a single 140 mg dose of evolocumab subcutaneously on Day 1.
- Evolocumab 140 mg - Total: Participants received a single 140 mg dose of evolocumab subcutaneously on Day 1.
Arm/Group | Evolocumab 140 mg - Normal Renal Function | Evolocumab 140 mg - Severe RI | Evolocumab 140 mg - ESRD Requiring Hemodialysis | Evolocumab 140 mg - Total
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/6 | 1/18
Other Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 2/6 | 4/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab 140 mg - Normal Renal Function (N=6) | Evolocumab 140 mg - Severe RI (N=6) | Evolocumab 140 mg - ESRD Requiring Hemodialysis (N=6) | Evolocumab 140 mg - Total (N=18)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Evolocumab 140 mg - Normal Renal Function (N=6) | Evolocumab 140 mg - Severe RI (N=6) | Evolocumab 140 mg - ESRD Requiring Hemodialysis (N=6) | Evolocumab 140 mg - Total (N=18)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.